CLINICAL TRIAL: NCT02620215
Title: Cervical Ripening Balloon in Induction of Labour at Term (CRBII) - A Prospective Randomized Controlled Trial
Brief Title: Cervical Ripening Balloon in Induction of Labour at Term
Acronym: CRBII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Tagore Shephali, Senior Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/2730
Record Dates: First submitted 2015-11-09; First posted 2015-12-02 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Pregnancy
MeSH Terms: interventions — KLK15 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical Ripening Balloon (Experimental): Cook® Cervical Ripening Balloon with Stylet Order number G19891 Reference Part Number J-CRBS-184000 Catheter (Fr) 18.0 Length (cm) 40 Balloon Volume (mL) 80
  Interventions: Device: Cervical Ripening Balloon
- Prostin (Active Comparator): Prostin E2 vaginal tablets contain the active ingredient dinoprostone, which is a naturally occuring female hormone also known as prostaglandin E2. Prostaglandins are involved in naturally starting labour. Dose of Prostin is 3 mg vaginally.
  Interventions: Drug: Prostin

INTERVENTIONS:
Device: Cervical Ripening Balloon — Cook® Cervical Ripening Balloon with Stylet Order number G19891 Reference Part Number J-CRBS-184000 Catheter (Fr) 18.0 Length (cm) 40 Balloon Volume (mL) 80
  Arms: Cervical Ripening Balloon
Drug: Prostin — Prostin E2 vaginal tablets contain the active ingredient dinoprostone, which is a naturally occuring female hormone also known as prostaglandin E2. Prostaglandins are involved in naturally starting labour. Dose of Prostin is 3 mg vaginally.
  Other Names: Prostin E2 vaginal tablets
  Arms: Prostin

SUMMARY:
About 1 in 6 deliveries in KKH are induced with prostaglandins. Inpatient induction can be a lengthy process especially when cervical priming is required. Although mechanical method of induction of labour (IOL) is established, its use in Singapore is uncommon. Systematic reviews comparing mechanical method against pharmacological and surgical IOL showed that mechanical method has similar efficacy with lower risk profile. As IOL is a common obstetric procedure, a revisit on the techniques is warranted. A multi-centre randomised controlled trial concluded that both cervical ripening balloon and prostaglandin are effective and complementary methods for IOL in uncomplicated singleton pregnancies, but did not examined the effects of pain.

The investigators propose to evaluate the adverse events in the 12 hours after CRB or 1st prostaglandin insertion, its efficiency in term singleton IOL in Singapore context and test the acceptability of women in Singapore in using the CRB as an alternative method of induction of labour while using a non-incremental balloon filling regime. Currently, there is no efficient method of induction that can be used safely in an outpatient setting. Through this study, the investigators hope to show that there are no major adverse events in the 12h after patients are induced with CRB, this potentially supports outpatient IOL with CRB which can reduce hospitalisation and medical costs. A non-incremental balloon filling regime will decrease time delays and may increase patient satisfaction during its use in induction of labour.

DETAILED DESCRIPTION:
This is a prospective cohort randomised controlled trial conducted at the KK Women's and Children's Hospital (KKH) and University Malaya Medical Centre (UMMC).

NICE guidelines on induction of labour defined uterine hyperstimulation as contractions more than 5 in 10 mins for more then 20 mins or contractions lasting more than 2 mins in duration. A retrospective study involving prostaglandin induction of labour showed that hyperstimulation occurred in 5.8% of cases. The sample size is calculated based on a 4.8% reduction in hyperstimulation in all induction of labour by CRB. At a level of significance of 5%, 80% power, 200 patients in each arm is required. Preliminary study by Tan TL et al had a dropout rate of 4.6%. Hence the proposed sample size is 420.

The investigators plan to collaborate on a multi-centre trial with the University Malaya Medical Centre. In which, each centre will recruit 210 patients for the study.

Randomization of the participants is achieved with third party sealed envelope allocation. 210 envelopes containing CRB allocation and another 210 identical envelopes containing prostin allocation will be prepared by a third party. The 420 envelops will be shuffled according to a computer randomisation code after sealing and labelled with a randomization allocation number from 1 to 420. The 210 envelops will then be handed to the each centre's PI, and will be kept in the clinical store on labour ward together with the stock of CRB and prostin.

Unfortunately, it is not possible to blind the allocation to the investigator or the patient. The investigator however has no part in observing any adverse events, the CTGs should be interpreted by the attending clinician and vet by team to avoid missing abnormal CTG. The patient herself will have to report contractions and pain scores and satisfaction scores with validated standard pain and satisfaction assessment tools to minimise the potential bias. The allocation will also be omitted from the database so as to blind the analyst in order to prevent manipulation.

There will be no additional clinic visit or labour ward admission required by the study. The potential patient receiving subsidized obstetric care who require elective IOL at term will be will be identified by doctors and clinical research coordinator in the subsidized clinic or labour ward or obstetric subsidized wards, and screened accordingly with inclusion criteria and exclusion criteria.

Inclusion criteria: Pregnant women aged 21 - 40 years old, singleton pregnancy, no major fetal anomaly, planned induction of labour at 37+0 weeks to 41+6 weeks gestation, vaginal delivery is appropriate, patient able to give informed consent to participate in the trial

Exclusion criteria: Spontaneous labour at start of planned induction, Bishop score <6 and cervical dilatation >=3 cm at start of induction, confirmed rupture of membrane, abnormal CTG at start of induction, caesarean section delivery is indicated, scarred uterus such as previous caesarean section, malpresentation in labour, patient withdraw consent to participate in the trial. Latex allergy, severe asthma and glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 21 - 40 years old
* Singleton pregnancy with no major fetal anomaly
* Planned induction of labour at 37+0 weeks to 41+6 weeks gestation
* Vaginal delivery is appropriate
* Patient able to give informed consent to participate in the trial

Exclusion Criteria:

* Spontaneous labour at start of planned induction
* Bishop score <6 and cervical dilatation >=3 cm at start of induction
* Confirmed rupture of membrane
* Abnormal CTG at start of induction
* Caesarean section delivery is indicated
* Scarred uterus such as previous caesarean section
* Malpresentation in labour
* Latex allergy, severe asthma and glaucoma
* Patient withdraw consent to participate in the trial

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 417 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Adverse events in the first 12 hours after Cook's Cervical Ripening Balloon insertion for induction of labour, in comparison to 1st prostin insertion | Up to 24 hours after induction of labour

SECONDARY OUTCOMES:
Efficacy of Cook's Cervical Ripening Balloonas a devide for induction of labour, in comparison to prostin, in achieving vaginal deliveries | Up to 96 hours after delivery
Patient satisfaction of the Cook's Cervical Ripening Balloon as a devide for induction of labour, in comparison to prostin, by using a 10-point scale | From induction of labour to up to 4 days after delivery
  Score 1 for poor and score 10 for excellent
Patients' experience of the Cook's Cervical Ripening Balloon as a devide for induction of labour, in comparison to prostin, by using a 10-point pain assessment scale | From induction of labour to up to 4 days after delivery
  Score 1 for no pain, score 3 for pain similar insertion of IV access line, and score 8 for labour pain at time of request for epidural or labour if no epidural is used

CONTACTS AND LOCATIONS:
Overall Officials: Shephali Tagore, MRCOG, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Grace Ng YH, Aminuddin AA, Tan TL, Kuppusamy R, Tagore S, Yeo GSH. Multicentre randomised controlled trial comparing the safety in the first 12 h, efficacy and maternal satisfaction of a double balloon catheter and prostaglandin pessary for induction of labour. Arch Gynecol Obstet. 2022 Jan;305(1):11-18. doi: 10.1007/s00404-021-06090-y. Epub 2021 May 11. PMID 33973051